CLINICAL TRIAL: NCT04645381
Title: Bone Erosions in Rheumatoid Arthritis - Characterization Evaluated by Imaging and Histology
Acronym: BERA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 675-897-002
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; High-resolution peripheral quantitative computed tomography; Radiography; Micro computed tomography; Histology
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Bone samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with RA

SUMMARY:
The aim of this study is to describe macro- and micro anatomical structures, including investigating vessels running in osseous pores in finger joints from participants with rheumatoid arthritis (RA) using histology and different imaging modalities. The perspectives are to increase understanding of the macro- and micro anatomic basis for bone erosions in RA, and possibly to provide new insights to the monitoring of patients with RA.

DETAILED DESCRIPTION:
This study is a descriptive, cross-sectional pilot study. The trial subjects will have their hands imaged by conventional radiography. The 2nd and 3rd digit metacarpophalangeal (MCP) joint will be scanned by high-resolution peripheral quantitative computed tomography (HR-pQCT). Patients with RA (n = 10) will be included and bone samples from MCP joints analyzed using microcomputed tomography (µCT) and histology.

ELIGIBILITY CRITERIA

Inclusion criteria:

* Age > 18 years.
* Participants diagnosed with RA according to the ACR/EULAR (2010) classification criteria or American Rheumatism Association 1987 revised criteria for the patients who were diagnosed before 2010.
* Indication for prosthesis surgery with total joint replacement of the MCP joint according to the clinical procedure (often radiological signs of osteoarthrosis (OA) in the MCP joint, joint pain, angular deformity and/or impairment of daily functions).

ELIGIBILITY:
RA Participants:

Inclusion Criteria:

* Age > 18 years
* Participants diagnosed with RA according to the ACR/EULAR (2010) classification criteria or American Rheumatism Association 1987 revised criteria for the patients who were diagnosed before 2010.
* Indication for prosthesis surgery with total joint replacement of the MCP joint according to the clinical procedure (often radiological signs of OA in the MCP joint, joint pain, angular deformity and/or impairment of daily functions).

Exclusion Criteria:

* Unable to give written informed consent.
* Active malignant disease, hypercalcemia, poor kidney function (estimated glomerular filtration rate < 35 mL/min), untreated hypo-/hyperthyroidism, pregnancy or wish thereof, previously fracture/dislocation of the investigated joint or metal prosthesis in joints of the investigated hand.

Bone sample will be excluded from analysis, if the following is present:

- Bone not adequate for analysis (fractured bone samples).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RA are recruited in conjunction with a routine visit at the Department of Orthopedic Surgery at Aarhus University Hospital or at the Regional Hospital Holstebro for assessment of surgical indication for joint replacement surgery on MCP joints by a specialist in orthopedic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Transcortical vessels and pores. | within 24 weeks after inclusion
  To identify and describe transcortical vessels and pores at the bare area in MCP joints from RA patients and describe the location, number, and compare intra- and extra-articularly by histology, μCT, and HR-pQCT.

SECONDARY OUTCOMES:
The bare area | within 24 weeks after inclusion
  To identify and describe the bare area in MCP joints from RA patients macroscopically, with imaging (HR-pQCT, conventional X-ray, μCT), and histology.
Bone erosions | within 24 weeks after inclusion
  To identify bone erosions by conventional X-ray, μCT, and HR-pQCT and assess inflammatory infiltrates using histology in RA patients.

OTHER OUTCOMES:
Microarchitecture | within 24 weeks after inclusion
  Microarchitecture in the cortical and trabecular bone compartment by HR-pQCT and μCT in RA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen-Margrethe Hauge, Professor, Study Director — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Central Region of Denmark
  - Regional Hospital Holstebro, Holstebro, Central Region of Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Therkildsen J, Klose-Jensen R, Langdahl B, Bruel A, Thomsen JS, Moger C, Stilling M, Keller KK, Hauge EM. Mapping the bare area and transcortical pores in finger joints: co-location with bone erosions in rheumatoid arthritis. RMD Open. 2026 Jan 22;12(1):e006371. doi: 10.1136/rmdopen-2025-006371. PMID 41571324